CLINICAL TRIAL: NCT01092325
Title: A Phase I/IIa Dose-Escalation Study Evaluating the Safety and Tolerability of CXL-1020 and Specific Effects on Electrocardiographic and Non-Invasive Hemodynamic Parameters in Patients With Chronic Heart Failure
Brief Title: Safety and Hemodynamic Effects and Pharmacokinetics of CXL-1020 in Patients With Stable Heart Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Cardioxyl Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CXL-1020-01
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1 CXL-1020 (Experimental): An intravenous infusion of CXL-1020 administered for a total of 4 hours over a total of 3 occasions separated by at least one week. Each of the 3 doses of CXL-1020 are different, starting with the lowest dose and increasing to the highest dose.
  Interventions: Drug: CXL-1020
- Cohort 1 Placebo (Placebo Comparator): A 4 hour infusion of Placebo administered one time randomly among the 3 active doses of CXL-1020 in cohort 1
  Interventions: Drug: Placebo for CXL-1020 Cohort 1
- Cohort 2 CXL-1020 (Experimental): An intravenous infusion of CXL-1020 administered for a total of 4 hours over a total of 3 occasions separated by at least one week. Each of the 3 doses of CXL-1020 are different, starting with the lowest dose and increasing to the highest dose.
  Interventions: Drug: CXL-1020
- Cohort 2 Placebo (Placebo Comparator): A 4 hour infusion of Placebo administered one time randomly among the 3 active doses of CXL-1020 in cohort 1
  Interventions: Drug: Placebo for CXL-1020 Cohort 2
- Echo Cohort A CXL-1020 (Active Comparator): A 4 hour infusion of a fixed dose of CXL-1020 which was studied in Cohort 1 or Cohort 2 which is expected to be well tolerated and have hemodynamic effect
  Interventions: Drug: CXL-1020 Dose for Echo Cohort A
- Echo Cohort B CXL-1020 (Active Comparator): CXL-1020 administered at a fixed rate for the initial 2 hours and at a higher fixed rate for the last 2 hours of a 4 hour infusion at doses which were studied in Cohort 1 or Cohort 2 and expected to be well tolerated and have hemodynamic effects
  Interventions: Drug: CXL-1020 Doses for Echo Cohort B

INTERVENTIONS:
Drug: CXL-1020 — Intravenous infusion of one of 3 active dosages of CXL-1020
  Arms: Cohort 1 CXL-1020
Drug: CXL-1020 — Intravenous infusion of one of 3 active dosages of CXL-1020 at dosages higher than in Cohort 1
  Arms: Cohort 2 CXL-1020
Drug: Placebo for CXL-1020 Cohort 1 — A 4 hour infusion of a IV solution containing 5% Dextrose in water (Sugar Water)
  Arms: Cohort 1 Placebo
Drug: Placebo for CXL-1020 Cohort 2 — A 4 hour infusion of a IV solution containing 5% Dextrose in water (Sugar Water)
  Arms: Cohort 2 Placebo
Drug: CXL-1020 Dose for Echo Cohort A — A 4 hour fixed dose of CXL-1020 which was studied in Cohort 1 or 2 which was demonstrated to be safe and well tolerated and have some anticipated hemodynamic effect
  Arms: Echo Cohort A CXL-1020
Drug: CXL-1020 Doses for Echo Cohort B — A 2 hour dose level of CXL-1020 which was studied in Cohort 1 or 2 which was demonstrated to be safe and well tolerated and have some anticipated hemodynamic effect followed by another higher 2 hour dose level of CXL-1020 which was studied in Cohort 1 or 2 which was demonstrated to be safe and well tolerated and have some anticipated hemodynamic effect
  Arms: Echo Cohort B CXL-1020

SUMMARY:
A Phase 1-2a Study of CXL-1020-01 in Patients with Stable Heart Failure

DETAILED DESCRIPTION:
This is a Phase I/IIa Dose-Escalation, First exposure in Humans, Study Evaluating the Safety and Tolerability of CXL-1020 and Specific Effects on Electrocardiographic and Non-Invasive Hemodynamic Parameters in Patients with Chronic Heart Failure. 4 weekly four-hour treatments involving ascending dosages of CXL-1020 with a randomly interspersed placebo dose within two or more unique patient cohorts. Separate echocardiography cohorts (Echo Cohort A and Echo Cohort B) will evaluate a sustained dose over 4 hours (ECHO A), and an ascending two dose level, 4-hour infusion (2 hours each) (ECHO B), in individual patients. Echo Cohort dosages will be determined from responses observed in previous cohort exposures.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for randomization, a patient MUST:

* Be a male or post menopausal or surgically sterile female outpatient between 18 and 85 years of age
* Have chronic Systolic HF due to primary/idiopathic dilated cardiomyopathy, coronary artery disease or hypertension, and stable for at least 30 days prior to screening
* Have a core echo lab confirmed left ventricular ejection fraction ≤ 40% in a baseline 2D-Echocardiogram prior to and within 60 days of the first dose of study medication with evidence of at least minimal LV dilation on the basis of an observed LV-EDV index that is above normal
* Have a baseline NT-Pro-BNP of greater than or equal to the top of the normal reference range (124pg/ml) prior to and within 60 days of the first dose of study medication
* Be on unchanging doses of HF medications (with exception of diuretic dosage) for 2 weeks prior to randomization without planned initiation of new hemodynamically active therapy during the conduct of the study
* Be capable of understanding the nature of the trial and be willing to participate as documented by written informed consent
* Be willing and able to comply with the study protocol requirements for the duration of the study, including pharmacokinetic sampling
* If a post-menopausal or surgically sterile female, confirmation of sterility status (Post menopausal or surgically sterile for at least 6 months) - (Post-menopausal subjects will require a urine pregnancy test for confirmation prior to enrollment and urine pregnancy tests prior to each dosing)
* If a fertile male, must be using 2 approved contraceptive methods (a condom and a spermicidal agent, even if the partner is using birth control) for the duration of the study and for 3 months following participation in the study and further agree to not donate sperm for 3 months after participation in the study. Must have a negative urine test for drugs of abuse and a negative ethanol breath test at screening and before each dosing period
* Have required local lab data within non-exclusionary ranges before each dosing

Exclusion Criteria:

In order to be eligible for randomization, a patient MUST NOT:

* Have participated in any investigational drug study within 30 days preceding randomization or have previously received therapy with CXL-1020
* Have a heart rate <50 or ≥ 90 BPM at baseline prior to randomization.
* Have a blood pressure >150 Systolic and/or >90 diastolic mmHg at baseline prior to randomization
* Have a systolic blood pressure of less than 100 mmHg at baseline prior to randomization
* Have QT/QTc prolongation > 460 msec or > 500msec in patients with preexisting bundle branch block (only applies to non-paced patients in sinus rhythm)
* Have experienced a documented symptomatic or electrocardiographically recorded episode of atrial fibrillation/flutter within 60 days before screening and be in normal sinus rhythm at each baseline before study drug is administered
* Have a history of sustained or hemodynamically significant VT or VF requiring cardioversion, or self-terminating VT associated with hypotension
* Have non-sustained VT (HR > 120 bpm) of 10 beats or more during monitoring in the baseline monitoring period prior to each dose of study medication, or in any Holter or EKG recording within 1 year of first dose of study medication.
* Have a weight or height that exceeds the specifications for the ICG Device of (greater than 341 pounds or taller than 7 feet 2 inches.)
* Be post-successful cardiac resuscitation
* Have a history of worsening HF within 30 days prior to screening as defined by:

  * Unscheduled ER or clinic visits relating to HF or hospital admission for management of HF
  * Treatment with intravenous inotropic or vasodilator drugs
* Be diagnosed with acute coronary syndrome or acute myocardial infarction within three months prior to screening
* Have a history of stroke (CVA) or transient ischemic attack (TIA) within six months prior to screening
* Have a history of CCS Class III or IV angina
* Be a patient whose HF etiology is attributable to either restrictive/obstructive cardiomyopathy, idiopathic hypertrophic cardiomyopathy (as defined by any wall thickness > 1.8 cm) or uncorrected severe valvular disease
* Be receiving concomitant therapy with any antiarrhythmic drugs other than amiodarone
* Have experienced the firing of an implantable ICD for documented ventricular ectopy within three months prior to screening
* Have a known allergy to the ICG Device sensor gel or adhesive
* Have unsuitable Echocardiographic Windows for the comprehensive Echo assessments required in the Echo cohorts (exclusion for echo cohorts only)
* Have a skin lesion at the site of the ICG Device sensor placement.
* Have a screening or baseline serum Na < 130 mEq/l or > 145 mEq/l; a serum K < 3.5 mEq/l or > 5.0 mEq/l; a serum Ca < 7.5 mg/dl or > 10 mg/dl; or a serum Mg < 1.6 mEq/l or > 3.0 mEq/l., or a digoxin level above 1ng/ml
* Have a screening TSH < 0.1 mcU/ml or > 5.0 mcU/ml
* Have a screening or baseline serum creatinine > 2.5 mg/dl; an ALT or AST >3 times the upper normal limit; or a hemoglobin < 10 g/dl
* Have taken ethanol within 24 hours or a PDE5 inhibitor within 96 hours of study admission
* Have other clinically significant laboratory or medical conditions that, in the opinion of the Investigator, make the patient unsuitable for evaluation in the study
* Have a generalized atopic state or a history of a mild to moderate documented drug allergy
* Be receiving a drug which is expected to possess the potential for a clinically significant pharmacokinetic interaction with CXL-1020, as defined in the IDB.

Note: Patients receiving cardiac resynchronization therapy for HF are eligible provided that the device has been placed for greater than 30 days and pacemaker settings can be left unchanged for the study period.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | From initial exposure to 30 days following exposure
  Safety is measured by assessment of multiple parameters including standard laboratory safety, changes in blood pressure and heart rate, changes in electrocardiogram, monitoring of heart rhythm via holter monitor, measurement of cardiac safety biomarkers such as plasma troponin as well as treatment emergent adverse events

SECONDARY OUTCOMES:
Hemodynamic Effects as Measured by Impedance Cardiography and Echocardiography | before during and following the infusion of study medication
  Standard measurement of impedance cardiography parameters will be made non invasively in all study cohorts. Echocardiography will be evaluated in parallel with Impedance cardiography in the Echo Cohorts
Plasma and Urinary Pharmacokinetics | From start of infusion until 18 hours post infusion
  Measurement of plasma samples and urine collections for CXL-1020 and metabolites. Samples are collected approximately 19 times from a intravenous catheter, before during and following infusion. In addition 4 collections of all freely voided urine will be collected from before infusion until 18 hours following infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Doug Cowart, Pharm D., Study Director — Cardioxyl Pharmaceuticals
Locations (1):
- Orange County Clinical Research Center, Tustin, California, United States

REFERENCES:
- [Result] A Phase I/IIa First in Man Safety and Tolerability Study of a Novel HNO Donor, CXL-1020, in Patients with Stable Congestive Heart Failure. Monday, April 4, 2011; 9:30 a.m. - 12:30 p.m., Ernest N. Morial Convention Center, Hall F; Poster Board #42
- [Derived] Sabbah HN, Tocchetti CG, Wang M, Daya S, Gupta RC, Tunin RS, Mazhari R, Takimoto E, Paolocci N, Cowart D, Colucci WS, Kass DA. Nitroxyl (HNO): A novel approach for the acute treatment of heart failure. Circ Heart Fail. 2013 Nov;6(6):1250-8. doi: 10.1161/CIRCHEARTFAILURE.113.000632. Epub 2013 Oct 9. PMID 24107588